CLINICAL TRIAL: NCT02544100
Title: Neonatal Neurologic Intensive Care Network of China
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xiamen Children's Hospital, Fujian of China (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Guangzhou Women and Children's Medical Center (Other); Yuying Children's Hospital of Wenzhou Medical University, Zhejiang of China (Unknown); Maternal and Child Health Hospital of Hubei Province (Other); The People's Hospital of Dehong Autonomous Prefecture (Other); Guangzhou Medical University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU5; NCT02606656 (obsolete NCT alias)
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Neonatal Encephalopathy; Suspected Neonatal Encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, Urine and CSF samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Database Entry / Biospecimen Collection: Systematic Medical information of infants born with severe encephalopathy entered into database. In addition, Blood, urine, CFS samples will be collected.
  Interventions: Other: Database Entry/Biospecimen Collection

INTERVENTIONS:
Other: Database Entry/Biospecimen Collection — blood, urine, CFS samples and medical data collected

SUMMARY:
The purpose of this study is to create a neonatal neurologic biological big data center named Neonatal Neurologic Intensive Care Network in China with neonatal systematic information, biological samples and genomics & genetic data on neonates born with neonatal severe encephalopathy. It also can predict brain injury as cerebral function monitoring through big data and recommend appropriate treatment. In addition, the following samples will be collected in a bio-bank in for future studies: blood, urine, and cerebrospinal fluid (CSF) samples.

DETAILED DESCRIPTION:
The purpose of this study is to create a neonatal neurologic biological big data center named Neonatal Neurologic Intensive Care Network in China with neonatal systematic information mainly including demographic, medical history, family condition, perinatal stage information, birth, growth & feeding status, imaging, biological samples and genomics & genetic data on neonates born with neonatal severe encephalopathy. It also can predict brain injury as cerebral function monitoring through big data and recommend appropriate treatment. There are seven children's hospitals from 6 provinces in China to join in the collaboration network in first recruiting. In addition, the following biological samples will be collected in a bio-bank for future studies: blood, urine, and cerebrospinal fluid (CSF) samples.

ELIGIBILITY:
Inclusion Criteria:

1. Postnatal age < or = 28 days
2. Written informed consent of parent or guardian

   With one of the following items
3. Hypoxic ischemic encephalopathy (HIE)
4. Hydrocephalus
5. Hypotonia
6. Interventricular hemorrhages
7. Intracranial calcifications
8. Intracranial hemorrhages
9. Meningitis and other brain infections
10. Metabolic diseases
11. Microcephaly
12. Neonatal stroke
13. Spina bifid
14. Cerebral arteriovenous malformations (AVMs)
15. Congenital brain malformations

Exclusion Criteria:

1. Known other major congenital anomalies but not not neurologic disease.
2. Failed to get sample or the volume of collected biosamples is not enough.
3. Parents refuse consent.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal with severe encephalopathy or suspected severe encephalopathy.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Blood Samples | In 72 hours
  Blood samples-based data of genetic and biomarkers for the monitoring of neonatal encephalopathy.
Number of Urine Samples | In 72 hours
  Urine samples-based data of biomarkers for the monitoring of neonatal encephalopathy.

SECONDARY OUTCOMES:
Number of Electronic Medical Records | To follow for the duration of hospital stay, an expected average of 4 weeks
  To collect systemic medical information about neonatal encephalopathy.
Neurodevelopment(Bayley Scores) | At the age of 18 months
  To evaluate neurodevelopmental function via Bayley Scores of Infant Development Mental Development Index (BSIDMI) and gain incidence of BSIMDI<70(Severe) or BSIMDI<85(Moderate).
Neurological Evaluation(GMFM-88 Scores) | At the age of 18 months
  To gain changes in standardized gross motor function using GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales, lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function).
Gene Mutation | At the age of 28 days
  To detect the mutation and characterize the genetic architecture and risk variants of neonatal malformation using different genomic methods.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Suarez JI, Geocadin R, Hall C, Le Roux PD, Smirnakis S, Wijman CA, Zaidat OO. The neurocritical care research network: NCRN. Neurocrit Care. 2012 Feb;16(1):29-34. doi: 10.1007/s12028-011-9612-x. PMID 21792751
- [Background] Narayanan JT, Murthy JM. New-onset acute symptomatic seizure in a neurological intensive care unit. Neurol India. 2007 Apr-Jun;55(2):136-40. doi: 10.4103/0028-3886.32784. PMID 17558117
- [Background] Hall CE, Mirski M, Palesch YY, Diringer MN, Qureshi AI, Robertson CS, Geocadin R, Wijman CA, Le Roux PD, Suarez JI; First Neurocritical Care Research Conference Investigators. Clinical trial design in the neurocritical care unit. Neurocrit Care. 2012 Feb;16(1):6-19. doi: 10.1007/s12028-011-9608-6. PMID 21792753
- [Background] Riviello JJ Jr. Pediatric neurocritical care. Introduction. Semin Pediatr Neurol. 2014 Dec;21(4):239-40. doi: 10.1016/j.spen.2014.12.009. Epub 2014 Dec 19. No abstract available. PMID 25727504
- [Background] Riviello JJ Jr, Chang C. The practice of pediatric neurocritical care by the child neurologist. Semin Pediatr Neurol. 2014 Dec;21(4):299-302. doi: 10.1016/j.spen.2014.12.007. Epub 2014 Dec 13. PMID 25727512
- [Background] Wainwright MS, Grimason M, Goldstein J, Smith CM, Amlie-Lefond C, Revivo G, Noah ZL, Harris ZL, Epstein LG. Building a pediatric neurocritical care program: a multidisciplinary approach to clinical practice and education from the intensive care unit to the outpatient clinic. Semin Pediatr Neurol. 2014 Dec;21(4):248-54. doi: 10.1016/j.spen.2014.10.006. Epub 2014 Nov 1. PMID 25727506
- [Background] Murphy SA, Bell MJ, Clark ME, Whalen MJ, Noviski N. Pediatric Neurocritical Care: A Short Survey of Current Perceptions and Practices. Neurocrit Care. 2015 Oct;23(2):149-58. doi: 10.1007/s12028-015-0120-2. PMID 25693892
- [Background] LaRovere KL, Graham RJ, Tasker RC; Pediatric Critical Nervous System Program (pCNSp). Pediatric neurocritical care: a neurology consultation model and implication for education and training. Pediatr Neurol. 2013 Mar;48(3):206-11. doi: 10.1016/j.pediatrneurol.2012.12.006. PMID 23419471
- [Background] Bonifacio SL, Glass HC, Peloquin S, Ferriero DM. A new neurological focus in neonatal intensive care. Nat Rev Neurol. 2011 Aug 2;7(9):485-94. doi: 10.1038/nrneurol.2011.119. PMID 21808297
- [Derived] Liu L, Xu SH, Zhang P, Lu CM, Cheng GQ. [Effect of red blood cell transfusion on the oxygenation of mesenteric tissue in premature infants]. Zhonghua Er Ke Za Zhi. 2018 Sep 2;56(9):680-685. doi: 10.3760/cma.j.issn.0578-1310.2018.09.009. Chinese. PMID 30180407